CLINICAL TRIAL: NCT03625492
Title: Effect of Potentially Irritating Beverages on Overactive Bladder Symptoms
Brief Title: Fluids Affecting Bladder Urgency and Lower Urinary Symptoms
Acronym: FABULUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other); Arbor Research Collaborative for Health (Other)
Responsible Party: Principal Investigator, Janis Miller, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00148419
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Overactive Bladder; Urinary Urgency; Urinary Bladder, Overactive; Urinary Incontinence, Urge; Caffeine; Alcohol Drinking; Lower Urinary Tract Symptoms
Keywords: artificial sweeteners; caffeine; alcohol drinking; urinary urgency; overactive bladder; urinary incontinence, urge; lower urinary tract symptoms
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Alcohol Drinking; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduce Potentially Irritating Beverages (Experimental): This group will receive a 7 minute video teaching participants to replace beverages that include caffeine, alcohol, artificial sweeteners, or acidic juices with equal volume intake of water, milk, or other beverages that do not have these ingredients in them.
  Interventions: Behavioral: Reducing Potentially Irritating Beverages
- Adopt Healthy Eating Habits (Active Comparator): This group will receive a 7 minute video teaching them the USDA guidelines for healthy eating.
  Interventions: Behavioral: Adopting the USDA Healthy Eating Habits

INTERVENTIONS:
Behavioral: Reducing Potentially Irritating Beverages — This group will receive a 7 minute video teaching participants to replace beverages that include caffeine, alcohol, artificial sweeteners, or acidic juices with equal volume intake of water, milk, or other beverages that do not have these ingredients in them.
  Arms: Reduce Potentially Irritating Beverages
Behavioral: Adopting the USDA Healthy Eating Habits — This group will receive a 7 minute video teaching them the USDA guidelines for healthy eating.
  Arms: Adopt Healthy Eating Habits

SUMMARY:
This study evaluates whether eliminating certain ingredients (caffeine, alcohol, artificial sweeteners, acidic juices) consumed in beverages reduces bladder symptoms of urinary frequency and urgency. Women with overactive bladder will be recruited. Half of these women will receive instructions to replace beverages containing these ingredients with beverages such as water or milk. The other half of participants will receive instructions on following the United States Department of Agriculture guidelines on healthy eating.

DETAILED DESCRIPTION:
It is commonly believed that it is better for women's bladders if intake of certain beverages is eliminated. Advice is given to women with frequency/urgency symptoms to avoid coffee or tea, sodas or pop, or any other drinks that contain alcohol, caffeine, artificial sweeteners or high acidic content. Although the investigators do not know the direct cause and effect of consuming beverages with these ingredients, there might be reduction in "irritating" sensation to toilet often because of urgency if the beverages with these ingredients are replaced by "non-irritating" beverages.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Daily intake of at least 16 oz. of potentially irritating beverages, defined as drinks that are caffeinated, artificially sweetened, citric/acidic, or alcoholic beverages
* Daily intake of at least 32 oz. of total beverages
* At least two of the following three qualifications: urinating greater than on average seven times during waking hours on 3-day diary, urinating routinely more than two times at night, answering "yes" to experiencing frequent, strong feelings of urgency to empty the bladder.

Exclusion Criteria:

* Men
* History of diabetes, spinal cord injury, multiple sclerosis, muscular dystrophy, cerebral palsy, dementia or Alzheimer's or stroke
* Currently pregnant or within one year of delivery
* Currently report symptoms of pain with urination or frequent urinary tract infections
* Uses diuretic medications, currently taking medication prescribed for bladder symptoms or have had surgery for incontinence with the last 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Urination frequency on 3-day bladder diary | 2-weeks
  Average number of times urinated per day on 3-day bladder diary

SECONDARY OUTCOMES:
Volume of urine per toileting event | 2-weeks
  Average volume of urine per day with each toileting event on 3-day bladder diary
Daily urination urgency symptoms (Adapted from Bower et al 2001) | 2-weeks
  The adapted question reads, "Typically, when you needed to go to the bathroom today you could…" with the five potential responses ranging from "make the urge go away" to "already feel the urine coming out." Urgency will be measured as the mean reported score for each three-day time period for the perception of bladder fullness questionnaires.
Perception of bladder fullness relative to urination delay ability (DeWachter, 2003) | 2-weeks
  On 3-day diary, participants will be asked to indicate their perception of bladder fullness when they urinated that day: "no bladder sensation," "urinating could easily be delayed for more than 30-60 minutes," "urinating could only be delayed for 30 minutes," "urinating could only be delayed for 5 minutes" and "immediate urinating will be mandatory and/or fear of leakage."
Bother associated with bladder symptoms (Coyne 2002) | 2-months
  The investigators will use only the "bother" questions of this larger Questionnaire about bladder symptoms. We modified the original think-back period of 4-weeks to instead think back to "the past 3 days" to characterize the bother of bladder symptoms under the varying conditions of each specific intervention period. Bother will be measured on the final day on the bottom of each of the 3-day diaries.
Urination frequency on 3-day diary (longer-term effect) | 2-months
  Average number of times urinated per day on 3-day bladder diary

CONTACTS AND LOCATIONS:
Overall Officials: Janis M Miller, PhD, Principal Investigator — University of Michigan; Megan O Schimpf, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Bower WF, Moore KH, Adams RD. A pilot study of the home application of transcutaneous neuromodulation in children with urgency or urge incontinence. J Urol. 2001 Dec;166(6):2420-2. PMID 11696802
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- [Background] De Wachter S, Wyndaele JJ. Frequency-volume charts: a tool to evaluate bladder sensation. Neurourol Urodyn. 2003;22(7):638-42. doi: 10.1002/nau.10160. PMID 14595606